CLINICAL TRIAL: NCT00617045
Title: Duloxetine in the Treatment of Postpartum-onset and Non-Postpartum Onset Major Depressive Disorder
Brief Title: Duloxetine for the Treatment of Postpartum Depression
Acronym: DuloxPPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor patient recruitment
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Kimberly Yonkers, Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC0609001827-Lilly-Duloxetine; F1J-US-X043 (Other Grant/Funding Number: Eli Lilly Pharmaceutical)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Postpartum Depression; Major Depressive Disorder
Keywords: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): type of experimental agent
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — Total treatment period is 12 weeks
  30mg po qd times 1 week
  60mg po qd times 11 weeks
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to assess whether the antidepressant, duloxetine, is equally effective as a treatment for subjects who have a Postpartum Onset Depression compared to subjects who have an onset of Major Depressive Disorder prior to delivery. The hypothesis is that duloxetine will be as effective in subjects with Postpartum Major Depressive Disorder as in subjects with a Major Depressive Disorder.

DETAILED DESCRIPTION:
Study was terminated because of poor enrollment

ELIGIBILITY:
Inclusion Criteria:

* adult female subjects age 18 and above if onset of depression within 4 weeks of delivery,or onset of depression antenatally either during pregnancy or before pregnancy
* must score greater than or equal to 12 on the Edinburgh Postnatal Depression Scale
* speak English or Spanish
* have access to a telephone
* provide written and verbal consent

Exclusion Criteria:

* have current or lifetime psychosis
* an unstable medical condition
* hypertension
* narrow-angle glaucoma
* liver disease
* seizure disorders
* bulimia
* anorexia
* mania
* substance abuse disorders
* have a known hypersensitivity to duloxetine or any of the active ingredients
* are in need of inpatient hospital treatment with an excluded medication
* adolescents under the age of 18

Medication Exclusion

* other antidepressants
* antipsychotic agents
* quinolone antibiotics
* Type 1C antiarrhythmics
* daily benzodiazepines
* Treatment with a monoamine oxidase inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in depression severity compared to baseline scores on the IDS-C between the two subject groups. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Yonkers, MD, Principal Investigator — Yale University
Locations (1):
- Perinatal & Postpartum Research Program 142 Temple ST Suite 301, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No